CLINICAL TRIAL: NCT07230743
Title: Comparison of Anxiety During Mask Induction of Anesthesia in Pediatric Patients With an Immersive/Interactive Technological Intervention Versus Traditional Care: A Latin American Experience
Brief Title: The Study Evaluates the Effect of an Interactive Projector as a Distraction for Children During Anesthetic Induction. The Primary Objective is to Reduce Perioperative Anxiety, Measured With the Modified Yale Preoperative Anxiety Scale (mYPAS).
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Alemana de Santiago (Other)
Collaborators: Universidad del Desarrollo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID 1483
Record Dates: First submitted 2025-09-08; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Anxiety After Surgery; Induction of Anesthesia; Anxiety Preoperative; Anesthesia Care; Technology Use; Child Anxiety
Keywords: Custom Projector-based Software Game; Pediatric Mask Induction Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group superiority trial with 1:1 individual randomization to BERT (a non-pharmacologic audiovisual projection during anesthetic induction) or usual care without BERT. The randomization sequence is created and implemented in REDCap, and group assignment remains concealed until setup in the operating room. The study is open-label-families and clinical staff can tell whether the projection is used-while data analysis is performed by team members who are not involved in delivering the intervention.
  Enrollment takes place at a single site (Ambulatory Pediatric Surgery Unit, Clínica Alemana de Santiago, Chile). Eligible participants are children 2-6 years scheduled for elective adenotonsillar surgery under general anesthesia. A caregiver is present in both arms. Outcomes are collected during induction on Day 0; caregivers are contacted again 14 days after surgery to complete the PHBQ-AS.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants, caregivers, and clinical staff (anesthesia/OR teams) are not masked. Outcome assessors who score mYPAS, HRAD+/-, and ICC from video recordings are masked to group assignment: recordings are framed to exclude any view of the projection/screen and audio cues are removed; raters receive only a study ID and time point. The data team/statistical analysts remain masked until the analysis plan is finalized and the database is locked. The allocation sequence is concealed within REDCap and is revealed to implementers only at the time of induction. Unmasking of raters or analysts will occur only for prespecified safety reviews or after database lock. Inter-rater agreement (intraclass correlation) will be monitored to ensure the quality of masked assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Parent-Present Induction (PPI) (Active Comparator): Participants in the Standard PPI group will undergo routine mask induction of anesthesia accompanied by a parent, with no additional structured distraction.
  Interventions: Other: Standard Parent-Present Induction (PPI)
- Technology Intervention group (Experimental): Participants in the Technology Intervention group will receive the same parent-present induction, with the addition of a custom projector-based video game intervention (BERT; Stanford Chariot Program, Palo Alto, CA). The interactive audiovisual content is displayed on a large projection screen strategically placed at the foot of the operating table to ensure optimal visibility for the pediatric patient. Children will be instructed to watch and engage with the content as they enter the operating room and throughout the induction process.
  Interventions: Device: Custom projector-based video game intervention (BERT; Stanford Chariot Program, Palo Alto, CA); Other: Standard Parent-Present Induction (PPI)

INTERVENTIONS:
Device: Custom projector-based video game intervention (BERT; Stanford Chariot Program, Palo Alto, CA) — The interactive audiovisual content is displayed on a large projection screen strategically placed at the foot of the operating table to ensure optimal visibility for the pediatric patient. Children will be instructed to watch and engage with the content as they enter the operating room and throughout the induction process.
  The intervention is designed to promote engagement and reduce perioperative anxiety. Research assistants will set up and operate the projection system and ensure appropriate timing and delivery. Caregivers and OR personnel will be permitted to interact with the child as usual during induction. The video intervention concludes upon loss of consciousness, at which point standard perioperative care resumes.
  Other Names: BERT
  Arms: Technology Intervention group
Other: Standard Parent-Present Induction (PPI) — Participants in the Standard PPI group will undergo routine mask induction of anesthesia accompanied by a parent, with no additional structured distraction.

SUMMARY:
This study is designed to evaluate the effect of technology as a distraction technique during anesthetic induction in children, starting from their arrival to the operating room. An interactive film will be displayed using a projector (BERT: Bedside Entertaining and Relaxation Tool) mounted on a whiteboard in front of the child's gurney. The primary outcome is perioperative anxiety, measured with the Modified Yale Preoperative Anxiety Scale (mYPAS).

DETAILED DESCRIPTION:
This study is a randomized, controlled, open-label, parallel-assignment clinical trial designed to evaluate the effect of a non-pharmacologic technological intervention (projected video game) on perioperative anxiety in children during anesthetic induction.

Study type: Prospective, comparative clinical trial. Randomization: Simple randomization in a 1:1 ratio using an electronic sequence generated and administered in REDCap®.

Masking: Open-label (no blinding), as healthcare staff, caregivers, and patients can identify the presence or absence of the projected video game during induction. However, statistical analyses will be performed by investigators who did not take part in the intervention's implementation, in order to minimize bias.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective procedures under general anesthesia at Clinica Alemana
* Parent or caregiver presence for mask induction
* ASA I, II
* Ages 2-6 years of age
* Spanish speaking
* Parental consent/patient assent

Exclusion Criteria:

* Patient or parental does not consent
* ASA ≥ III
* Emergency surgery
* Intravenous induction of anesthesia
* Patient with a significant neurological condition or major developmental disability
* Severe visual or auditory defects
* Patients admitted using a crib as the mode of transport

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pediatric anxiety | Perioperative/anesthetic induction
  Pediatric anxiety levels during mask induction as measured through the Modified Yale Preoperative Anxiety Scale (mYPAS). The Modified Yale Preoperative Anxiety Scale (mYPAS) is a 22-item checklist divided into five categories: "activity," "vocalization," "emotional expressiveness," "apparent arousal," and "relationship with parents." Each category consists of a list of interrelated behaviors, the most representative of which is the score for that category. The mYPAS score ranges from 23.3 to 100; the threshold for considering patients with anxiety is > 30.

SECONDARY OUTCOMES:
Affect and Cooperation | Perioperative/anesthetic induction
  To measure patient affect and cooperation during mask induction, measured by HRAD +/- scale. The Happy, Relaxed, Anxious, Distressed with a yes/no measure of cooperation (HRAD ±) is an observational affect scale developed to clinically assess affect and cooperation during inhalational induction and minor procedures.
Compliance | Perioperative/anesthetic induction
  To measure cooperation and compliance during mask induction, with the ICC (Induction Compliance Checklist). This scale contains a list of 11 behaviors that the child may exhibit when the face mask is placed near them during induction. The score ranges from 0 to 10, with 0 indicating that the child cooperates and shows no mask-rejecting behaviors, and 10 indicating the worst expected response. The higher the score on the ICC scale, the greater the child's rejection of the surgical mask. The authors recommended that a score of 6 or higher be considered traumatic anesthesia.
Caregiver Satisfaction With the Induction Experience | Perioperative/after anesthetic induction
  To assess caregiver satisfaction regarding the projector-based software program for mask induction, measured by Parent Satisfaction Survey. This survey consists of a score from 0 to 5; from 0 = very unsatisfied to 5 = very satisfied.
Long-term behavioral outcomes | 2 weeks after surgery
  To measure incidence of postoperative behavioral outcomes after anesthesia event, measured by Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS). The PHBQ is comprised of 27 items among six subscales (general anxiety and regression, separation anxiety, eating disturbance, aggression toward authority, apathy/withdrawal, anxiety about sleep). This method produces a possible range of scores from 27 - 135 (with with higher scores, worse outcomes).
Correlation to HRAD+/- to mYPAS | Single time point at mask application during anesthetic induction (Day 0, intraoperative)
  To measure correlation of HRAD+/- to mYPAS
Correlation to HRAD+/- to ICC | Single time point at mask application during anesthetic induction (Day 0, intraoperative).
  To measure correlation of the cooperation component of HRAD+/- to ICC

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Alemana de Santiago, Vitacura, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Given the pediatric, single-center design and small sample size, the risk of re-identification remains non-trivial even after de-identification. In addition, our consent forms do not explicitly authorize external IPD sharing. We will share aggregate numerical results only (e.g., group means, SDs, effect sizes, confidence intervals) in publications and on ClinicalTrials.gov, and provide the protocol and SAP upon request.

REFERENCES:
- [Background] Jenkins BN, Kain ZN, Kaplan SH, Stevenson RS, Mayes LC, Guadarrama J, Fortier MA. Revisiting a measure of child postoperative recovery: development of the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery. Paediatr Anaesth. 2015 Jul;25(7):738-45. doi: 10.1111/pan.12678. Epub 2015 May 9. PMID 25958978
- [Background] Rodriguez ST, Jang O, Hernandez JM, George AJ, Caruso TJ, Simons LE. Varying screen size for passive video distraction during induction of anesthesia in low-risk children: A pilot randomized controlled trial. Paediatr Anaesth. 2019 Jun;29(6):648-655. doi: 10.1111/pan.13636. Epub 2019 Apr 14. PMID 30916447
- [Background] Fefferman MS, Fraser AE, Takemoto CM, Menendez A, Graetz TJ, Beres AL. Prospective, observational validation of HRAD±, a novel pediatric affect and cooperation scale. Paediatric Anaesthesia. 2024;34(4):376-384.
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Jerez-Molina C, Lázaro-Alcay JJ, Ullán-de la Fuente AM. Adaptación transcultural al español de la Induction Compliance Checklist para evaluar el comportamiento infantil durante la inducción anestésica. Enfermería Clínica (English Edition). 2017;27(5):271-276.
- [Background] Jerez C, Ullan AM, Lazaro JJ. Reliability and validity of the Spanish version of the modified Yale Preoperative Anxiety Scale. Rev Esp Anestesiol Reanim. 2016 Jun-Jul;63(6):320-6. doi: 10.1016/j.redar.2015.09.006. Epub 2015 Nov 26. English, Spanish. PMID 26633606
- [Background] Yun R, Caruso TJ. Identification and Treatment of Pediatric Perioperative Anxiety. Anesthesiology. 2024 Nov 1;141(5):973-983. doi: 10.1097/ALN.0000000000005105. No abstract available. PMID 39163600
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Vieco-Garcia A, Lopez-Picado A, Fuentes M, Francisco-Gonzalez L, Joyanes B, Soto C, Garcia de la Aldea A, Gonzalez-Perrino C, Aleo E. Comparison of different scales for the evaluation of anxiety and compliance with anesthetic induction in children undergoing scheduled major outpatient surgery. Perioper Med (Lond). 2021 Dec 14;10(1):58. doi: 10.1186/s13741-021-00228-x. PMID 34903293